CLINICAL TRIAL: NCT03875755
Title: Reduction of Insulin Therapy Under Myo-inositol for the Treatment of Gestational Diabetes Mellitus: a Randomized Multicenter and Prospective Trial. MYO-GDM Study
Brief Title: Myo-inositol for Reduction of Insulin Therapy in Gestational Diabetes Mellitus
Acronym: MYO-GDM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160940J
Record Dates: First submitted 2019-01-25; First posted 2019-03-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Diabetes; Pregnancy; MYO-INOSITOL; Oral supplementation
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myo Inositol (Experimental): The women will receive 2 caps of Myo Inositol with acid folic a day, until delivery
  Interventions: Dietary Supplement: Myo Inositol
- Placebo (Placebo Comparator): The women will receive 2 caps of placebo (acid folic) a day, until delivery
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Myo Inositol — One soft gel capsule containing MI 600 mg and folic acid 200 μg twice a day, until delivery.
  Other Names: INOFOLIC
  Arms: Myo Inositol
Other: Placebo — One soft gel capsule of placebo (folic acid 200 μg) twice a day until delivery.
  Arms: Placebo

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as hyperglycemia first-diagnosed during pregnancy. Glycemic control reduces GDM-related complications. With the new diagnostic criteria of GDM, up to 25% of pregnant women have GDM, whereas it was previously 6-10% in France. Therefore caring for women with GDM is very time-consuming. Therapeutic strategy includes dietary and lifestyle measures and additional insulin therapy for 15 to 40% of the women with GDM if the glycemic targets are not achieved after a period of 1 to 2 weeks of diet. Insulin therapy is imperfect for the following main reasons: need for education (i.e. subcutaneous administration, dose titration), hypoglycemia and weight gain, limited acceptance and high cost. Psychosocial deprivation is associated with more cases of GDM and health accessibility may be unequal.

MYO-INOSITOL (MI) is an oral dietary supplement, which reduces insulin resistance. Women with GDM are deficient in MI. MI supplementation safely prevents GDM by 65 to 87% in high-risk women. A pilot study has shown a 75% reduction of the need for insulin during GDM not controlled by diet.

The coordinator investigator propose here, for the first time, a randomized controlled study evaluating MI versus placebo in women with newly diagnosed GDM.

DETAILED DESCRIPTION:
Prospective, multicenter, superiority, randomised, double blind study with two arms.

1. In the 23 participating centers selection of women with GDM between 6 to 37 (+6 days) amenorrhea weeks
2. Explanation of protocol, with signature of consent in case of acceptation.
3. Randomization

   * Experimental group: The women will receive 2 caps of MI with acid folic a day, until delivery
   * Control group: The women will receive 2 caps of placebo (containing only acid folic) a day, until delivery

   In both arms, the participants will be routinely followed up during pregnancy:
   * diet education,
   * self-monitoring of blood glucose before and after meals
   * and during follow-up insulin therapy if glucose value targets are unmet
4. Routine monitoring of the women with GDM in both arms, up to delivery, without use of other oral hypoglycemic agents during pregnancy.

   At delivery:
   * MI (or placebo) will be stopped
   * Events during pregnancy will be collected
5. Last visit three months after delivery. Oral glucose tolerance test, anthropometric measures for women and their child.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Singleton pregnancy
* GDM diagnosed during pregnancy according to IADPSG (International Association of the Diabetes and Pregnancy Study Groups) criteria, i.e.

  * fasting plasma glucose between 92 mg/dL (5.1 mmol/L) and 125 mg/dL (6.9 mmol/L)
  * and/or 1-hour plasma glucose value after 75 g oral glucose tolerance test (OGTT) ≥ 180 mg/dL (10.0 mmol/L)
  * and/or 2-hour plasma glucose value between 153 mg/dL (8.5 mmol/L) and 199 mg/dL ((11.0 mmol/L)
* or overt diabetes according to 2-hours post OGTT plasma glucose value ≥ 200 mg/dl
* 6 to 37 (+6 days) amenorrhea weeks at the time of randomization
* Capacity for self-monitoring of blood glucose
* Signed informed consent

Exclusion Criteria:

* Insulin use before randomization during this pregnancy
* Use of other oral hypoglycemic agents during this pregnancy
* Long time corticosteroid treatment
* Pre-existing diabetes before pregnancy
* Overt diabetes diagnosed during pregnancy according to fasting plasma glucose ≥ 126 mg/dL (7 mmol/l)
* Lack of Social Insurance
* Insufficient French understanding and speaking
* Participant in another investigational drug study at inclusion visit
* Fetal malformation diagnosed by previous fetal ultrasound
* Personal history of any bariatric surgery
* Hypersensitivity to any ingredient of dietary supplement formulation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The participants in this study are pregnant women with gestational diabetes mellitus.
Enrollment: 1080 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Rate of patients requiring insulin therapy during pregnancy | At any time during pregnancy up to delivery; assessed up to 29 weeks.
  Rate of patients requiring insulin therapy (either basal or prandial). .

SECONDARY OUTCOMES:
- Rate of patients requiring basal insulin therapy during pregnancy- /Rate of patients requiring prandial insulin therapy during pregnancy | At any time during pregnancy up to delivery; assessed up to 29 weeks.
  This information will be retrieved from the glucose meter, and if not available, from the woman's diary
- Doses of basal and prandial insulin at delivery- Gestation age when insulin is began - Duration of insulin treatment | At delivery; assessed up to 29 weeks.
  * Dose of basal insulin (UI) at delivery, if any
  * Dose of prandial insulin (UI) at delivery, if any
  * Gestational age (SA) when basal insulin is started.
  * Gestational age (SA) when prandial insulin is started
  * Duration of basal insulin treatment at delivery, if any
  * Duration of prandial insulin treatment at delivery, if any
Gestational weight gain | At any time during pregnancy up to delivery; assessed up to 29 weeks.
  * Gestational weight gain (Kg) during pregnancy
  * Gestational weight gain (Kg) between inclusion and delivery
Hypoglycemia | from randomization to delivery; assessed up to 29 weeks.
  * Severe hypoglycemia: requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions. Plasma Glucose concentrations may not be available during an event, but neurological recovery following the return of plasma/capillary glucose to normal is considered sufficient evidence that the event was induced by a low plasma/capillary glucose concentration.
  * Documented symptomatic hypoglycemia: event during which typical symptoms of hypoglycemia are accompanied by a measured capillary glucose concentration <70 mg/dL (<3.9 mmol/L).
  * Asymptomatic hypoglycemia: event not accompanied by typical symptoms of hypoglycemia but with a measured capillary glucose concentration <60 mg/dL (<3.3 mmol/L).
Capillary glucose levels | From the beginning of MI Supplementation to delivery;assessed up to 29 weeks.
  The women will be asked to perform 6 measures a day. Capillary glucose values will be retrieved from the glucose meter, and if not available, from the woman's diary.
Neonatal complications | At delivery; assessed up to 29 weeks
  * Birth weight ≥ 4000g; ≥ 4500g ; large and small for gestational age infant
  * Neonatal hypoglycemia defined as at least a blood glucose value lower than 2.0 mmol/l after 2 hours of life during the two first days of life if the newborn is asymptomatic
  * Shoulder dystocia, defined as vaginal cephalic delivery
  * Birth injury defined as plexus injury or clavicle fracture
  * Preterm delivery:
  * Late preterm infant (between 32 and 37 completed amenorrhea weeks)
  * Very preterm infant (28-31 completed amenorrhea weeks)
  * Extreme preterm infant (less than 28 completed amenorrhea weeks)
  * Low Apgar score: 5-min Apgar score < 7• Jaundice, defined as need for neonatal phototherapy • Neonatal respiratory distress syndrome, based on the clinical course, chest X-ray finding, blood gas and acid-base values • Medical need for admission to pediatric or neonatal intensive care unit during the three days following birth • Malformations: the types of malformation will be recorded.
Preeclampsia - Pregnancy-induced hypertension - Cesarean section - Maternal inpatient admission during pregnancy | At any time during pregnancy up to delivery; assessed up to 29 weeks.
  * Preeclampsia (blood pressure ≥ 140/90 mmHg on two measurements four hours apart and proteinuria of at least 300 mg/24 hours or 3+ or more on dipstick testing or proteinuria/creatinuria >30 in a random urine sample)
  * Pregnancy-induced hypertension: in women with no known hypertension before pregnancy, blood pressure ≥ 140/90 mmHg on two measurements four hours apart without proteinuria and having needed to begin anti-hypertensive therapy
  * Maternal inpatient admission during pregnancy after inclusion, not including hospitalization just after delivery
Side effects | From the beginning of MI Supplementation to delivery; assessed up to 29 weeks.
  The investigators expect MI not to have any side effect at the dose 1200 mg/day, but possible side effects will be collected.
Results of oral glucose tolerance test | 3 months after delivery
  Test will be performed by the women 3 months post partum
Infant anthropometrics. | At month 1, month 2 and month 3
  These data will be collected from children's health record
Acceptance/satisfaction of 2 strategies: score | At delivery; assessed up to 29 weeks.
  Evaluation of the patient's satisfaction about their treatment for GDM at delivery : give a score of 0 to 100: 0 not satisfied; 100 totally satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COSSON, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Avicenne, Bobigny
  - Hopital Avicenne, Bobigny

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Croze ML, Soulage CO. Potential role and therapeutic interests of myo-inositol in metabolic diseases. Biochimie. 2013 Oct;95(10):1811-27. doi: 10.1016/j.biochi.2013.05.011. Epub 2013 Jun 10. PMID 23764390
- [Background] Unfer V, Carlomagno G, Dante G, Facchinetti F. Effects of myo-inositol in women with PCOS: a systematic review of randomized controlled trials. Gynecol Endocrinol. 2012 Jul;28(7):509-15. doi: 10.3109/09513590.2011.650660. Epub 2012 Feb 1. PMID 22296306
- [Background] Corrado F, D'Anna R, Di Vieste G, Giordano D, Pintaudi B, Santamaria A, Di Benedetto A. The effect of myoinositol supplementation on insulin resistance in patients with gestational diabetes. Diabet Med. 2011 Aug;28(8):972-5. doi: 10.1111/j.1464-5491.2011.03284.x. PMID 21414183
- [Background] D'Anna R, Di Benedetto V, Rizzo P, Raffone E, Interdonato ML, Corrado F, Di Benedetto A. Myo-inositol may prevent gestational diabetes in PCOS women. Gynecol Endocrinol. 2012 Jun;28(6):440-2. doi: 10.3109/09513590.2011.633665. Epub 2011 Nov 28. PMID 22122627
- [Background] Matarrelli B, Vitacolonna E, D'Angelo M, Pavone G, Mattei PA, Liberati M, Celentano C. Effect of dietary myo-inositol supplementation in pregnancy on the incidence of maternal gestational diabetes mellitus and fetal outcomes: a randomized controlled trial. J Matern Fetal Neonatal Med. 2013 Jul;26(10):967-72. doi: 10.3109/14767058.2013.766691. Epub 2013 Mar 1. PMID 23327487
- [Background] D'Anna R, Scilipoti A, Giordano D, Caruso C, Cannata ML, Interdonato ML, Corrado F, Di Benedetto A. myo-Inositol supplementation and onset of gestational diabetes mellitus in pregnant women with a family history of type 2 diabetes: a prospective, randomized, placebo-controlled study. Diabetes Care. 2013 Apr;36(4):854-7. doi: 10.2337/dc12-1371. Epub 2013 Jan 22. PMID 23340885
- [Background] D'Anna R, Di Benedetto A, Scilipoti A, Santamaria A, Interdonato ML, Petrella E, Neri I, Pintaudi B, Corrado F, Facchinetti F. Myo-inositol Supplementation for Prevention of Gestational Diabetes in Obese Pregnant Women: A Randomized Controlled Trial. Obstet Gynecol. 2015 Aug;126(2):310-315. doi: 10.1097/AOG.0000000000000958. PMID 26241420
- [Background] Lubin V, Shojai R, Darmon P, Cosson E. A pilot study of gestational diabetes mellitus not controlled by diet alone: First-line medical treatment with myoinositol may limit the need for insulin. Diabetes Metab. 2016 Jun;42(3):192-5. doi: 10.1016/j.diabet.2016.01.005. PMID 26948394